CLINICAL TRIAL: NCT01366651
Title: An Open-Label Study to Evaluate the Penetration of Doripenem in Cerebrospinal Fluid After Doripenem Administration in Pediatric Subjects Less Than 1 Year Chronological Age
Brief Title: A Study of Doripenem in CerebrospinalFluid After Doripenem Administration in Pediatric Patients Less Than 1 Year of Age
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Trial terminated early per business decision.
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CR016189; DORIPED1002 (Other: Janssen Research & Development, LLC); 2011-001114-33 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2011-04-14; First posted 2011-06-06 (Estimated); Last update posted 2013-12-06 (Estimated); Status verified 2013-12

CONDITIONS: Meningitis
Keywords: Doripenem; DORIPED1002; Intravenous; Pediatric; Antibiotic; Meningitis
MeSH Terms: conditions — Meningitis | interventions — Doripenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Doripenem (Experimental): Doripenem Type=exact number unit=mg/kg number=10 form=solution for injection route=intravenous use every 8 hours for 2 days (total of 5 doses) for patients <12 weeks of age.Doripenem 500-mg sterile powder will be supplied for the study in single use glass vials.,Doripenem Type=exact number unit=mg/kg number=30 form=solution for injection route=intravenous use every 8 hours for 2 days (total of 5 doses) for patients 12 weeks to <1 year of age. Doripenem 500-mg sterile powder will be supplied for the study in single use glass vials.
  Interventions: Drug: Doripenem

INTERVENTIONS:
Drug: Doripenem — Type=exact number, unit=mg/kg, number=30, form=solution for injection, route=intravenous use, every 8 hours for 2 days (total of 5 doses) for patients 12 weeks to <1 year of age.
Drug: Doripenem — Type=exact number, unit=mg/kg, number=10, form=solution for injection, route=intravenous use, every 8 hours for 2 days (total of 5 doses) for patients <12 weeks of age.

SUMMARY:
The purpose of this study is to characterize the penetration of doripenem in the cerebral spinal fluid in pediatric patients <1 year of age who are hospitalized and have a documented or suspected infection and are planning to, or undergoing treatment with intravenous (IV) antibiotics.

DETAILED DESCRIPTION:
This is a multicenter, open-label (identity of treatment is known to patient's parent/legal guardian/caregiver and to all study staff) study to characterize the penetration of doripenem in the cerebral spinal fluid (CSF) in pediatric patients <1 year of age who are hospitalized but medically stable, and who have a documented or suspected infection and are planning to, or undergoing treatment with antibiotics administered intravenously (in a vein, abbreviated as "IV"). Doripenem will not replace the patients' prescribed antibiotic(s). The study includes 3 phases: a pretreatment phase consisting of an up to 24-hour screening period; a 2-day open-label treatment period when doripenem will be administered, and CSF and blood samples will be collected, and a follow-up visit approximately 1 week after administration of the last dose of doripenem. The total duration of the study is approximately 10 days. During the study, patients <12 weeks of age will receive a 10 mg/kg doripenem 1-hour IV infusion via a central or peripheral venous line (a catheter inserted in a large vein) every 8 hours; patients 12 weeks to <1 year of age will receive a 30 mg/kg doripenem 1-hour IV infusion every 8 hours. A total of 5 doses of doripenem will be administered over a 2-day period while the patient is in the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patient is expected to require hospitalization for the entire open-label phase of the study.
* Patient must be scheduled to have cerebral spinal fluid obtained via a lumbar puncture (referred to as a "spinal tap") or ventriculoperitoneal (VP) shunt tap within 3 days of enrollment into this study.
* Patient must have documented or suspected infection and is planning to, or undergoing treatment with IV antibiotics.
* Parent or the patient's legally acceptable representative must have signed an informed consent document indicating they understand the purpose of and procedures required for the study and are willing to allow the infant to participate in the study.

Exclusion Criteria:

* Clinically significant abnormal values for hematology or clinical chemistry at screening that, at the option of the investigator, are not consistent with the patient's underlying disease(s) or therapies.
* Any condition at screening that, in the opinion of the investigator, may interfere with the assessments of this study.
* Patients with substantially compromised renal (kidney) function: e.g., urine output is <0.25cc/kg/hr within the 24 hours before screening.
* History of clinically significant allergies to medications, especially known hypersensitivity or intolerance to carbapenems, penicillins, or other Beta-lactam antibiotics.
* Known allergy to heparin or history of heparin-induced thrombocytopenia, if an in-dwelling cannula (e.g., heparin lock) or central line is used.
* Patients concomitantly treated with or having received imipenem/cilastin within 48 hours before study drug administration.
* Patients concomitantly treated with probenecid or valproic acid (VPA).

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2012-03; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Doripenem concentrations in CSF and plasma | For up to 2 days

SECONDARY OUTCOMES:
Number of patients with adverse events | Up to Day 9
Changes in clinical laboratory test results | From Day -1 to Day 9
Changes in physical examination results reported as adverse events | From Day -1 to Day 9
Changes in vital signs measurements | From Day -1 to Day 9
Changes in concomitant therapy | From Day -1 to Day 9
The number of patients with changes from baseline in clinical laboratory test results | From Day -1 to Day 9
The number of patients who receive concomitant therapy | From Day -1 to Day 9

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Development, L.L.C., Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Leuven, Belgium

REFERENCES:
- See also: An Open-Label Study to Evaluate the Penetration of Doripenem in Cerebrospinal Fluid After Doripenem Administration in Pediatric Subjects Less Than 1 Year Chronological Age — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=6&filename=CR016189_CSR.pdf